CLINICAL TRIAL: NCT06868576
Title: Progestin-Primed Ovarian Stimulation Versus Gonadotrophin-Releasing Hormone Antagonist for Patients Undergoing Assisted Reproductive Technology: a Randomized Clinical Trial
Brief Title: PPOS Protocol Versus GnRH Anatagonist for Expected Normal Responder Patients Undergoing ART : a Randomized Clinical Trial
Acronym: PPOS vs GnRH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Hassan Badawy Gadallah, Dr, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD-10-2023
Record Dates: First submitted 2025-02-18; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: PPOS; GnRH Antagonist; Assisted Reproductive Techniques
MeSH Terms: interventions — Dydrogesterone; cetrorelix

STUDY DESIGN:
Intervention Model Description: Three hundred twenty-eight women will be divided into 2 groups (A and B), each group will consist of 164 patients:
  *Group A (Study group): Includes 164 patients that will undergo progestin primed ovarian stimulation (PPOS) protocol using dydrogesterone.
  *Group B (control group): Includes 164 patients that will receive the conventional GnRH antagonist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patients that will undergo progestin primed ovarian stimulation (PPOS) protocol using dydrogesterone (Experimental)
  Interventions: Drug: Dydrogesterone Oral Tablet
- patients that will receive the conventional GnRH antagonist. (Active Comparator)
  Interventions: Drug: Cetrorelix (Cetrotide)

INTERVENTIONS:
Drug: Dydrogesterone Oral Tablet — Dydrogesterone 20mg tablets daily in PPOS protocol in ovarian stimulation starting from day 2 or 3 of the menstrual cycle until the triggering day
  Arms: patients that will undergo progestin primed ovarian stimulation (PPOS) protocol using dydrogesterone
Drug: Cetrorelix (Cetrotide) — This will be the conventional antagonist in ovarian stimulation given from day 6 of the menstrual cycle until the triggering day
  Arms: patients that will receive the conventional GnRH antagonist.

SUMMARY:
The aim of this study is to compare the efficacy and safety of Progestin-Primed Ovarian Stimulation (PPOS) protocol versus the fixed GnRH antagonist protocol in expected normal responder patients undergoing intracytoplasmic sperm injection (ICSI) with frozen-thawed embryo transfer (FET). By evaluating key clinical outcomes, including ovarian response, embryological parameters, and pregnancy rates, this study seeks to determine the relative advantages and limitations of each protocol.

DETAILED DESCRIPTION:
In this prospective, non-inferiority trial, we will compare the efficacy and safety of the GnRH antagonist and PPOS protocols in 328 infertile women undergoing ICSI in Kasr Al-Ainy IVF department, Cairo University, Egypt. Before the trial, investigators were required to provide all information related to the clinical trial, including the possible benefits and risks, other therapeutic choices and the right to withdraw, via a written consent. After being provided with sufficient time to decide whether to participate and the opportunity to ask questions, all participants were required to provide written informed consent before study inclusion.

ELIGIBILITY:
Inclusion Criteria:

* • Women who had history of infertility for ≥1 year.

  * Women whose age <40 years old by the end of the study.
  * Anti-Mullerian hormone > 1.2 ng/ml.
  * Antral follicle count ≥ 5.

Exclusion Criteria:

* • Age ≥ 40 years old.

  * Women who are diagnosed as polycystic ovarian syndrome.
  * Women with endometriosis stage 3 or 4.
  * Documented previous IVF/ICSI cycles with no oocytes retrieved.
  * Women with contraindications to controlled ovarian stimulation.
  * Patients who refuse to share in the study.

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 328 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy | 7 weeks of gestational age
  The presence of fetal pulsations by ultrasound at 7 weeks of gestational age

SECONDARY OUTCOMES:
Incidence of moderate/severe OHSS | before triggering injection and within 9 days after triggering injection
Number of metaphase 2 oocytes | within 1 day of ovum pick up
number of 2 PN embryos | within 1 day of ovum pick up
Biochemical pregnancy | 2-3 weeks after embryo transfer
  Quantitative Beta chorinioic gonadotrophin (B-HCG) hormone levels in blood 2 to 3 weeks after embryo transfer.

CONTACTS AND LOCATIONS:
Locations (1):
- Ciro University Kasr Alainy OBGYN Hospital, Cairo, Alquahira, Egypt